CLINICAL TRIAL: NCT01342094
Title: A Double-masked Study of DE-111 Ophthalmic Solution Versus Timolol Ophthalmic Solution 0.5% in Patients With Primary Open Angle Glaucoma or Ocular Hypertension - Phase 3, Confirmatory Study -
Brief Title: DE-111 Against Timolol Ophthalmic Solution 0.5%
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01111005
Record Dates: First submitted 2011-04-24; First posted 2011-04-26 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-06

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: Primary open angle glaucoma or ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- DE-111 ophthalmic solution (Experimental): DE-111 ophthalmic solution (one drop at a time, once daily) and Placebo ophthalmic solution (one drop at a time, BID) in both eyes.
  Interventions: Drug: DE-111 ophthalmic solution; Drug: Placebo ophthalmic solution
- Timolol ophthalmic solution 0.5% (Active Comparator): Timolol ophthalmic solution 0.5% (one drop at a time, BID) and Placebo ophthalmic solution (one drop at a time, once daily) in both eyes.
  Interventions: Drug: Timolol ophthalmic solution 0.5%; Drug: Placebo ophthalmic solution

INTERVENTIONS:
Drug: DE-111 ophthalmic solution
  Arms: DE-111 ophthalmic solution
Drug: Timolol ophthalmic solution 0.5%
  Arms: Timolol ophthalmic solution 0.5%
Drug: Placebo ophthalmic solution

SUMMARY:
DE-111 ophthalmic solution will be evaluated for superiority in comparison with Timolol ophthalmic solution 0.5%, in IOP(intraocular pressure ) -lowering effect in primary open-angle glaucoma or ocular hypertension patients, in a multicenter, randomized, double-masked, parallel-group comparison study. Safety will be compared and evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary open angle glaucoma or ocular hypertension
* Provided signed, written informed consent
* 20 years of age and older
* If a subject is a female of childbearing potential, she must utilize reliable contraceptive throughout the study, and must have a negative urine pregnancy test prior to enrollment into this study

Exclusion Criteria:

* Females who are pregnant, nursing or planning a pregnancy, or females of childbearing potential who are not using a reliable method of contraception
* Presence of any abnormality or significant illness that could be expected to interfere with the study

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Santen study sites, Osaka, Osaka, Japan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to randomization all participants in the study were receiving Timolol ophthalmic solution 0.5% (one drop at a time, BID).
Groups:
- DE-111: DE-111 ophthalmic solution (one drop at a time, once daily) and Placebo ophthalmic solution (one drop at a time, BID) in both eyes.
- Timolol: Timolol ophthalmic solution 0.5% (one drop at a time, BID) and Placebo ophthalmic solution (one drop at a time, once daily) in both eyes.
Period: Overall Study
Arm/Group | DE-111 | Timolol
Started | 82 | 84
Completed | 77 | 81
Not Completed | 5 | 3
Not completed — Adverse Event | 5 | 0
Not completed — Not meeting inclusion/exclusion criteria | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Subjects who have instilled the investigational drug at least once.
Groups:
- Total: Total of all reporting groups
Arm/Group | DE-111 | Timolol | Total
Number analyzed (Participants) | 82 | 84 | 166
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 35 | 81
  >=65 years | 36 | 49 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (11.4) | 63.1 (12.4) | 62.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 46 | 90
  Male | 38 | 38 | 76
Region of Enrollment [Number; unit: participants]
  Japan | 82 | 84 | 166

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Diurnal IOP (Intraocular Pressure) at End of Study
Description: Mean diurnal IOP (intraocular pressure) was calculated as an average of IOP (intraocular pressure) at 9:30 (pre-dose), 11:30 and 17:30.
Time Frame: Week 0(Baseline) and Week 4(End of Study)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DE-111 | Timolol
Number analyzed (Participants) | 82 | 84
mmHg | -3.2 (2.1) | -1.7 (2.1)
Statistical Analysis 1: Comparison: DE-111 vs Timolol; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-2.2 to -0.9]

ADVERSE EVENTS:
Time Frame: Week 0(Baseline) and Week 4(End of Study)
Arm/Group | DE-111 | Timolol
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/84
Other Adverse Events (participants affected / at risk) | 11/82 | 2/84
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DE-111 (N=82) | Timolol (N=84)
Ocular hyperaemia (Eye disorders) | 6 | 1
Conjunctival hyperaemia (Eye disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No